CLINICAL TRIAL: NCT01666106
Title: Osteonecrosis of the Jaw (ONJ) Case Registry
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101102
Record Dates: First submitted 2012-06-22; First posted 2012-08-16 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Osteonecrosis of the Jaw

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with cancer and ONJ: Subjects with cancer and positively adjudicated ONJ

SUMMARY:
Osteonecrosis of the Jaw (ONJ) Case Registry

DETAILED DESCRIPTION:
The purpose of the ONJ case registry is to describe the natural history of positively-adjudicated ONJ in subjects with cancer with an observation period of 5 years. Most of these subjects are expected to have received bone antiresorptive agents such as bisphosphonates or denosumab together with cancer-specific therapies (eg, chemotherapy, steroids, or anti-angiogenics). It is also possible that the registry will include subjects with cancer who developed ONJ without exposure to any antiresorptive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) with diagnosis of cancer
* Newly diagnosed, positively-adjudicated ONJ
* ECOG <=2 and expected survival ≥3 months
* Willing to provide access to previous and future medical and dental information
* Subject or subject's legally acceptable representative has provided written informed consent

Exclusion Criteria:

* History of radiation to the jaws administered for the treatment of cancer
* Subject will not be available for protocol required study visits, to the best of the subject and investigator's knowledge.
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with cancer and ONJ
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Resolution rate and time to ONJ resolution | 5 years
  * Resolution: complete coverage of the exposed bone by mucosa in the absence of clinical symptoms
  * Improvement: a decrease in the stage or severity of the lesion
  * Progression: an increase in the stage or severity of the lesion
  * Stable: not resolved, improved, or progressed

SECONDARY OUTCOMES:
The clinical features of ONJ, including severity and staging at enrollment | 5 years
The frequency of risk factors for incident ONJ | 5 years
  Characterize the frequency of risk factors for incident ONJ such as a history of inflammatory dental disease (periodontal and dental abscesses), dentoalveolar procedures, smoking, use of antiangiogenic agents, and duration/dosing regimens of antiresorptive medications prior to the development of ONJ
Therapeutic treatment patterns for ONJ | 5 years
  Characterize treatment patterns of antiresorptive medications subsequent to incident ONJ such as the proportion of subjects who continue to be treated with antiresorptive medications by specific agents and ONJ severity and stage
Treatment patterns of antiresorptive agents subsequent to incident ONJ | 5 years
  Characterize subsequent treatment patterns for ONJ including antimicrobial oral rinses, antibiotics, and surgery

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (57):
- United States (20):
  - Research Site, Beverly Hills, California
  - Research Site, Duarte, California
  - Research Site, Denver, Colorado
  - Research Site, Farmington, Connecticut
  - Research Site, Stratford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Baltimore, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, Buffalo, New York
  - Research Site, Mineola, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
- Canada (5):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Québec, Quebec
- Denmark (2):
  - Research Site, Aarhus C
  - Research Site, København Ø
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Oulu
- France (5):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Saint-Herblain
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Mühlhausen
  - Research Site, München
  - Research Site, Regensburg
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Italy (5):
  - Research Site, Alessandria
  - Research Site, Brescia
  - Research Site, Lecce
  - Research Site, Roma
  - Research Site, Torino
- Spain (3):
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid
- United Kingdom (3):
  - Research Site, Cardiff
  - Research Site, London
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Schiodt M, Vadhan-Raj S, Chambers MS, Nicolatou-Galitis O, Politis C, Coropciuc R, Fedele S, Jandial D, Zhang J, Ma H, Saunders DP. A multicenter case registry study on medication-related osteonecrosis of the jaw in patients with advanced cancer. Support Care Cancer. 2018 Jun;26(6):1905-1915. doi: 10.1007/s00520-017-4003-2. Epub 2017 Dec 23. PMID 29275525
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com